CLINICAL TRIAL: NCT00970398
Title: Effect of Infant Formula With Bovine Milk Osteopontin on Infant Growth, Health and Immune functions-a Double-blind Randomized Trial
Brief Title: Effect of an Infant Formula on Infant Growth, Health and Immune Functions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biostime, Inc. (Industry)
Collaborators: Arla Foods (Industry); Children's Hospital of Fudan University (Other); University of California, Davis (Other); University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 200816609
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Health; Growth; Immune Functions
Keywords: Infant formula; Bovine milk Osteopontin; growth; health; immune functions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Reference group (No Intervention): Human milk breastfeeding
- Control formula (Active Comparator): Standard infant formula, with no Osteopontin supplemented.
  Interventions: Other: Standard infant formula
- Formula with 50% Osteopontin (Active Comparator): Infant formula supplemented with bovine milk Osteopontin at 50% level of that of breast milk.
  Interventions: Other: Infant formula supplemented with bovine milk Osteopontin
- Formula with 100% Osteopontin (Active Comparator): Infant formula supplemented with bovine milk Osteopontin at 100% level of that of breast milk.
  Interventions: Other: Infant formula supplemented with bovine milk Osteopontin

INTERVENTIONS:
Other: Infant formula supplemented with bovine milk Osteopontin — Infant formula supplemented with bovine milk osteopontin at 50% and 100% levels of that of breast milk respectively.
  Other Names: Lactopontin
  Arms: Formula with 100% Osteopontin; Formula with 50% Osteopontin
Other: Standard infant formula — Infant formula without supplementation of bovine milk Osteopontin
  Other Names: Lactopontin
  Arms: Control formula

SUMMARY:
The specific objectives of this study are to evaluate the effects of bovine milk osteopontin added to infant formula on infant growth, health and immune functions.

DETAILED DESCRIPTION:
Breast-fed infants will be used as a reference group and formula-fed infants will be fed control formula or the same formula supplemented with Osteopontin at a concentration 50% or 100% of that of breast milk. The hypothesis is that supplementation of bovine milk Osteopontin in infant formula will have positive effects on infant growth, health and immune functions.

ELIGIBILITY:
Mothers Inclusion Criteria:

* Healthy, 19-40 years of age
* Plan to exclusively breast-fed or formula-fed

Infants Exclusion Criteria:

* Gestational age < 37 or > 42 weeks
* Birth weight < 2.5kg or > 4 kg
* Having congenital diseases
* Having birth Asphyxia
* Having birth infections

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 320 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-09 (Actual); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Concentrations of immune cells and cytokines of IL-6, IL-10, and IL-12 in infant's blood samples will be measured to evaluate immune functions. | 1, 4, and 6 postnatal months

SECONDARY OUTCOMES:
Anthropometric parameters: body length, body weight, and head circumferences at each visit. | 1, 2, 3, 4, 5, and 6 postnatal months
Dietary, stool consistency and well being recorded by 3 day questionnaires | 1, 2, 3, 4, 5, and 6 postnatal months
Adverse events and concomitant medications recorded by heath forms as a measure of safety and tolerability. | 1, 2, 3, 4, 5, and 6 postnatal months

CONTACTS AND LOCATIONS:
Overall Officials: Yongmei Peng, M.D., Principal Investigator — Children's Hospital of Fudan University; Bo Lonnerdal, Ph.D., Principal Investigator — University of California, Davis
Locations (1):
- Children's Hospital of Fudan University, Shanghai, China

REFERENCES:
- [Background] Ashkar S, Weber GF, Panoutsakopoulou V, Sanchirico ME, Jansson M, Zawaideh S, Rittling SR, Denhardt DT, Glimcher MJ, Cantor H. Eta-1 (osteopontin): an early component of type-1 (cell-mediated) immunity. Science. 2000 Feb 4;287(5454):860-4. doi: 10.1126/science.287.5454.860. PMID 10657301
- [Background] Nagatomo T, Ohga S, Takada H, Nomura A, Hikino S, Imura M, Ohshima K, Hara T. Microarray analysis of human milk cells: persistent high expression of osteopontin during the lactation period. Clin Exp Immunol. 2004 Oct;138(1):47-53. doi: 10.1111/j.1365-2249.2004.02549.x. PMID 15373904
- [Background] Rollo EE, Hempson SJ, Bansal A, Tsao E, Habib I, Rittling SR, Denhardt DT, Mackow ER, Shaw RD. The cytokine osteopontin modulates the severity of rotavirus diarrhea. J Virol. 2005 Mar;79(6):3509-16. doi: 10.1128/JVI.79.6.3509-3516.2005. PMID 15731245
- [Derived] Lonnerdal B, Kvistgaard AS, Peerson JM, Donovan SM, Peng YM. Growth, Nutrition, and Cytokine Response of Breast-fed Infants and Infants Fed Formula With Added Bovine Osteopontin. J Pediatr Gastroenterol Nutr. 2016 Apr;62(4):650-7. doi: 10.1097/MPG.0000000000001005. PMID 26465791